CLINICAL TRIAL: NCT04158531
Title: Rational Extra-eloquent Closed-loop Cortical Stimulation (REC2Stim) as a Treatment for Refractory Epilepsy in the Primary Sensorimotor Cortex.
Brief Title: REC2Stim as a Treatment for Refractory Epilepsy in the Primary Sensorimotor Cortex.
Acronym: REC2Stim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Dorien van Blooijs, study coordinator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL66795.041.18; NEF17-07 (Other Grant/Funding Number: Dutch Epilepsy Foundation); METC19-336 (Registry Identifier: MREC Utrecht)
Record Dates: First submitted 2019-10-30; First posted 2019-11-08 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Epileptic Seizure; Epilepsy Intractable; Motor Seizure
Keywords: cortical electrical stimulation; seizure detection; network stimulation
MeSH Terms: conditions — Seizures; Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: This study is an early feasibility study in which the effect and safety of cortical network stimulation in patients with central lobe epilepsy is investigated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REC2Stim (Experimental): Use electrocorticography (ECoG)-based seizure detection and cortical network stimulation upon seizure onset detection.
  Interventions: Device: ECoG sensing and stimulation

INTERVENTIONS:
Device: ECoG sensing and stimulation — Implant electrodes and a sensing+stimulation device, and use this for suppression of seizure activity
  Other Names: Activa PC+S

SUMMARY:
People with central lobe epilepsy (CLE), with seizures arising from the primary sensorimotor cortex, typically show a high rate of convulsive seizures that do not respond to anti-epileptic drugs, but have a large impact on quality of life. They often seek surgical relief, but since the area contains the body's indispensable sensorimotor representation, CLE surgery will lead to permanent functional deficits. Cortical stimulation case studies in CLE have shown seizure frequency reduction of more than 90%, but in our experience, stimuli in the central lobe can hardly be applied without interfering with motor function.

The investigators propose cortical electrical stimulation therapy of a conceptually novel type. The investigators systematically determine individual stimulation settings, stimulation site and a seizure detection algorithm. In REC2Stim (Rational Extra-eloquent Closed-loop Cortical Stimulation), at the start of a seizure, a train of electric pulses is delivered to a nearby extra-eloquent area connected with the epileptogenic area within the sensorimotor cortex. Success will constitute a therapeutic modality for pharmaco-resistant patients with an epileptic focus in eloquent areas.

DETAILED DESCRIPTION:
The investigators will include ten patients with CLE, aged 16 years and older, in whom pre-surgical chronic intracranial EEG monitoring has revealed a seizure onset in the primary sensorimotor cortex. Patients should have on average at least two seizures per day.

Clinical intracranial EEG monitoring (normally 7-10 days) will be extended with two extra monitoring days, for systematic testing of different stimulation settings and their effect on interictal epileptiform EEG activity (as a surrogate marker for ictal epileptiform activity), from which site and parameters for chronic stimulation will be determined.

Upon removal of the clinically implanted electrodes, a neurostimulator with sensing capabilities, Activa PC+S, will be implanted and attached to two subdural leads with electrodes covering the predefined stimulation site and the eloquent epileptogenic area.

During a data collection phase, stimulation-free data will then be collected to train the seizure detection algorithm up to at least 50% sensitivity.

Finally, the REC2Stim phase will be started, in which cortical stimulation is applied when seizure activity is detected. Study participation is one year. When REC2Stim turns out effective in month 10 and 11 after implantation of the neurostimulator, 2 weeks of sham stimulation will follow in month 12.

ELIGIBILITY:
Inclusion Criteria:

* potential central lobe epilepsy
* on average 2 or more seizures per day or ongoing Epilepsia Partialis Continua (EPC)
* mentally and physically capable of giving informed consent
* minimally 3 anti-epileptic drugs been admitted without effect on seizure frequency (refractory epilepsy)

Exclusion Criteria:

* coagulopathy, including use of anticoagulant or antiplatelet agents
* known allergy to the materials of the implant
* progressive neurological or systemic disease
* contra-indications to the presence of a chronically implanted device, such as the need for repeated MRI, or concurrent infections
* any brain lesion that would place the patient at an elevated risk for bleeding
* any progressive brain disease, e.g. Rasmussen's encephalitis or glioma
* presence of any active implanted metallic device, such as cardiac pace-maker, vagal nerve or deep brain stimulator, cochlear implants, spinal cord stimulator or metallic parts from non-medical origin
* presence of aneurysm clips
* seizure onset zone (SOZ) outside eloquent cortex

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
seizure frequency - diary recorded in an app (MedApp) | study start until 1 year after implantation of last patient
  the number of seizures per day
seizure severity - diary recorded in an app (MedApp) | study start until 1 year after implantation of last patient
  the severity of the seizures, experienced by the patient. A scale of intensity from 0-10 (low - high severity) can be selected. Also the seizure type can be selected.

SECONDARY OUTCOMES:
Motoric functioning - muscle strength as part of neurological examination | study start until 1 year after implantation of last patient
  The investigators perform neurological examination during each outpatient clinic visit. We test muscle strength and scale that with the Medical Research Council Scale (MRC) (0-5: no contraction - normal strength).
Motoric functioning - coordination as part of neurological examination | study start until 1 year after implantation of last patient
  The investigators perform neurological examination during each outpatient clinic visit. Coordination is rated as normal or abnormal.
Motoric functioning - sensibility as part of neurological examination | study start until 1 year after implantation of last patient
  The investigators perform neurological examination during each outpatient clinic visit. Sensibility is rated as normal or abnormal.
Motoric functioning - reflexes as part of neurological examination | study start until 1 year after implantation of last patient
  The investigators perform neurological examination during each outpatient clinic visit. Reflexes are rated as normal or abnormal.
Simple functional abilities - nine hole peg test | study start until 1 year after implantation of last patient
  The investigators use the nine-hole peg test before implantation and 1 year after implantation. The investigators record the time it takes to place 9 sticks in openings and back on the plate again.
Complex functional abilities - Action Research Arm Test (ARAT) | study start until 1 year after implantation of last patient
  The investigators use the ARAT before implantation and 1 year after implantation. Scale ranges from 0-57 points (bad - normal performance).
Quality of life questionnaire | study start until 1 year after implantation of last patient
  The patient fills in the Assessment of Quality of Life (AQoL-8D). Scale ranges from 35-175 (high - low quality of life).
Participation abilities - Utrecht´s Scale for Evaluation of Rehabilitation (USER)- Participation questionnaire | study start until 1 year after implantation of last patient
  The patient fills in the USER-participation questionnaire. Score ranges from 0-500 (low - good participation)

CONTACTS AND LOCATIONS:
Overall Officials: Frans Leijten, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
selected datasets will be available through a public repository after publication of results
Time Frame: From January 2023, no end date